CLINICAL TRIAL: NCT01396343
Title: Environmental and Genetic Risk Factors for Pediatric Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: New York University (Other); Massachusetts General Hospital (Other); State University of New York at Buffalo (Other); University of Alabama at Birmingham (Other); Mayo Clinic (Other); Children's Hospital of Philadelphia (Other); Boston Children's Hospital (Other); Baylor College of Medicine (Other); Loma Linda University (Other); Children's Hospital Colorado (Other); University of Texas (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); Washington University School of Medicine (Other); Children's National Research Institute (Other); Primary Children's Hospital (Other); The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 5R01NS071463 (NIH)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Pediatric Multiple Sclerosis
Keywords: Pediatric Multiple Sclerosis; Relapsing Remitting Multiple Sclerosis; Clinically Isolated Syndrome; Demyelinating Disease
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Demyelinating Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Total 41ml sample: 17ml plasma/DNA, 10ml serum, 9ml lymphocytes and 5ml RNA frozen.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pediatric MS Case: Demographic and Medical History Questionnaire, Environmental Exposure Questionnaire, Food Frequency Questionnaire, Blood Sample Collection
- Pediatric Control: Demographic and Medical History Questionnaire, Environmental Exposure Questionnaire, Food Frequency Questionnaire, Blood Sample Collection

SUMMARY:
The purpose of this study is to better understand multiple sclerosis (MS) in children and adolescents, to learn if it differs from adult MS and to investigate if genes or environmental exposures or a combination of both put children and adolescents at risk for getting MS.

DETAILED DESCRIPTION:
The overall goal of this project is to determine whether well-established environmental and genetic risk factors for adult onset MS play an important role in susceptibility to pediatric-onset MS. Our study design is based on the hypothesis that genetic influences, specifically variation at HLA-DRB1 and other confirmed non-MHC MS loci, as well as environmental exposures including EBV infection and tobacco smoke, contribute to disease risk. In addition, we will also examine the relationship between serum levels of 25(OH) vitamin D3 and prior vitamin D status, and risk for pediatric onset MS. Finally, we will investigate whether specific G x E, and other multivariable relationships influencing risk exist for pediatric-onset MS. There are 16 collaborating sites other than UCSF that will enroll cases and controls for this study.

ELIGIBILITY:
Children are eligible for this study as cases if:

* They have MS or clinically isolated syndrome (CIS):

  * MS: As defined by the 2010 McDonald criteria for diagnosis of MS (Polman 2010),
  * CIS: A first demyelinating event indicating high risk for MS (i.e., one clinical event involving the spinal cord, the optic nerve, the brainstem or cerebellum, or occasionally the hemispheres) and at least 2 silent T2 bright areas on a brain or spinal cord MRI (at least one must be in the brain); AND
* They are three years of age or older; AND
* Disease onset occurred before 18 years of age.

Patients are not eligible for study participation if:

* Disease onset occurred more than 4 years prior to the opportunity to enroll; OR
* They have had an organ transplant; OR
* They are known to have neuromyelitis optica (NMO).

Children are not eligible to participate as pediatric controls if:

* They are two years of age or younger; OR
* They are 22 years of age or older; OR
* They are known to have MS or another demyelinating disease (for example, neuromyelitis optica or acute disseminated encephalomyelitis); OR
* They have a biological family member who has been enrolled as a control; OR
* They have an immediate, biological family member (parent/sibling) who has been diagnosed with MS; OR
* They have an autoimmune disorder (except asthma or eczema); OR
* They have had an organ transplant; OR
* They have a chronic neurological condition with major disability (this does not include, for example, migraine, controlled seizures, and mild learning disabilities such as ADD or ADHD).

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Case patients seen at the 16 participating Pediatric MS Center Clinics. Control patients seen at the Pediatric Clinics of the same institution as MS cases.
Sampling Method: Non-Probability Sample
Enrollment: 1276 (Actual)
Dates: Start 2011-10; Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Identify risk factors and their respective contribution to developing pediatric multiple sclerosis | 4 year data collection, 1 year analysis
  The primary objective of this study is to determine if risk factors identified for adult MS such as HLA-DRB1*1501/1503, EBV, 25(OH) vitamin D3 insufficiency, and exposure to cigarette smoking are also risk factors for pediatric MS, and if there are interactions between them analyzing data collected from questionnaires for environmental exposure, demographic and food frequency as well as sample blood specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle L Waubant, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (17):
- United States (17):
  - Center for pediatric-onset demyelinating diseases at the Children's Hospital of Alabama, Birmingham, Birmingham, Alabama
  - Pediatric MS Clinic, Children's Hospital, Loma Linda University, San Bernardino, California
  - UCSF Pediatric MS Center, San Francisco, California
  - Children's Hospital Colorado, University of Colorado School of Medicine, Aurora, Colorado
  - Pediatric MS Clinic, Children's National Medical Center, Washington D.C., District of Columbia
  - Pediatric MS Clinic, Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Partners Pediatric MS Center at the Massachusetts General Hospital for Children, Boston, Massachusetts
  - Pediatric MS Clinic, Children's Hospital Boston, Boston, Massachusetts
  - Regional Pediatric MS Center at Mayo Clinic, Rochester, Minnesota
  - Pediatric MS Clinic, Washington University School of Medicine, St Louis, Missouri
  - Pediatric MS Center of the Jacobs Neurological Institute, University of Buffalo, Buffalo, New York
  - New York University Langone Medical Center, New York, New York
  - The Cleveland Clinic, Cleveland, Ohio
  - Pediatric MS Clinic, Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pediatric MS Center, University of Texas, Southwestern Medical Center, Dallas, Texas
  - The Blue Bird Circle Clinic for MS at Texas Children's Hospital, Houston, Texas
  - Pediatric Neurology Clinic, Primary Children's Hospital, Salt Lake City, Utah